CLINICAL TRIAL: NCT01686490
Title: LifeSkills Video Training in Patients About to Receive an Automatic Implantable Cardioverter-Defibrillator
Brief Title: LifeSkills Video Training in Patients About to Receive an Automatic Implantable Cardioverter-Defibrillator (AICD)
Acronym: AICD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Williams LifeSkills (Industry)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Virginia P. Williams, Ph.D., President,, Williams LifeSkills
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2924526; 1R41HL083635-01A2 (NIH)
Record Dates: First submitted 2012-06-27; First posted 2012-09-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Focus Whether After Implant Pre-AICD Video Was Helpful
Keywords: AICD; focus groups; cognitive-behavioral video/workbook training; pre-implant concern/distress about upcoming AICD
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- D. (Other): The focus is evaluation of LifeSkills Video/Workbook for patients about to receive an AICD. Patients who now have received their AICD were given a video/workbook pre-implantation as an intervention to reduce their concerns/distress. After implantation, they will be asked what was and was not helpful about the materials they received.
  Interventions: Behavioral: Video/workbook for patients about to receive an AICD; Behavioral: LiveSkills Video/Workbook for patients about to receive an AICD

INTERVENTIONS:
Behavioral: Video/workbook for patients about to receive an AICD — will view the 3 completed sections of the video/workbook
Behavioral: LiveSkills Video/Workbook for patients about to receive an AICD — This exploratory intervention first met in a focus group with healthcare professionals and another focus group with patients who already had received an automatic implantable cardiac defibrillator to learn more about what video and accompanying workbook material it would be helpful for patients to receive pre-inplantation. Another focus group was held with post-implantation patients asking them what additional knowledge would have been helpful. Three sections of the video with accompanying workbook were then produced and given to pre-inplantation patients. A focus group was then held with these patients after their procedure to ask them what had and had not proved helpful.

SUMMARY:
The purpose of this trial was to develop the initial sections of a video/DVD cassette that provided guidance about mastering stressful situations for patients who had been informed that they need an implantable cardioverter-defibrillator (AICD). We adapted the existing LifeSkills video (which was already been shown effective in patients with heart diseases) to the specific needs of patients with AICD's. Before its development, we held separate focus groups with healthcare providers of AICD patients, pre-implantation patients, and post-implantation patients. After the video/accompanying workbook was produced, we held an additional focus group with patients who had received the video/workbook before receiving their AICD.

DETAILED DESCRIPTION:
Patients who had received the video/workbook told the focus group leader that they wanted more information about their AICD and a clearer presentation about how stress management was related to living with their AICD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age> 21 years old)
* For one of the initial focus groups and for the focus group of patients who had watched the produced modules: Patients who have received a recommendation for an AICD and have agreed to have it in the pre-implantation stage (do not already have the implant)
* For the other initial focus group: patients who already have an AICD.

Exclusion Criteria:

* Patients who are medically unstable [New York Heart Association class IV heart failure, recent (within 30 days) myocardial infarction or admission for unstable angina or worsening heart failure, in-patients, or patients who were admitted less than 1 month before potential enrollment will be excluded].
* Patients who are suffering from other medical illnesses: only the following categories will be exclusionary: Diseases that cause severe cognitive impairment that may lead to inability to understand or follow study procedures (i.e., severe dementia, identified by the patients' inability to repeat the study procedures and by a mini-mental status exam that will be done if dementia is suspected); Diseases that cause severe psychotic symptoms leading to disorientation (i.e., hepatic encephalopathy).
* Patients who are actively suicidal (suspected from the suicide question on the depression questionnaire
* Patients who cannot understand the study procedures due to cognitive or language barriers (provided an effort was made to offer translation).
* The process for dealing with individuals who indicate that they may be suicidal, depressed or anxious will be as follows: Immediately upon receipt of the completed questionnaires at the coordinating office, the Beck Depression Inventory and the Impact of Event Scale will be evaluated. If the responses indicate suicidal ideation the subject will be called and asked to contact his/her primary care provider for an immediate appointment. The primary care provider will be contacted that day to inform him/her of the finding. If the responses to the Impact of Event Scale or the BDI indicate stress or depression, a letter will be sent to the subject recommending that he/she contact the primary care provider. A copy of the letter will be forwarded to the PCP.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Whether patients understood the contents of the produced sections of the video/workbook and whether these contents were helpful. This will be determined by their comments during a focus group which will be held after they have watched the video. | After AICD patients who watched the video/workbook before implantation have been implanted.
  AICD patients who watched the first three sections of the proposed video with accompanying workbook will be asked in a focus group if they found the information comprehensible and if the information was helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gordon Rogers, MD, Principal Investigator — Duke University, Eed Director, Cardiac Transplant and Mechanical Circulatory Support Program
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States